CLINICAL TRIAL: NCT04887688
Title: Toward Smart Personalized Electrotherapy for Enhanced Healing of Ischemic Wounds
Brief Title: Exciflex for Chronic Wound Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F2166-R
Record Dates: First submitted 2021-04-16; First posted 2021-05-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Wound; Diabetes; Spinal Cord Injury; Ischemic Wound
MeSH Terms: conditions — Diabetes Mellitus; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: At the baseline assessment, the wound dressing will be removed and wound status will be evaluated. Participants will then be randomly assigned to the intervention group (Group A) or control group (Group B).
  Progressive changes in wound size, indicative of wound healing, will be determined using 3D digital stereophotogrammetry (LifeViz 3D system, Quantificare Inc., San Mateo, CA) together with wound swabs to collect wound bed fluid. The study cohort will comprise Veterans with ischemic wounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Wound treated using exciflex (Experimental): Intervention treated wounds in Group A participants will be covered using the exciflex bandage which will be activated to deliver ES using a 10% duty cycle, i.e. ES will be active for 1 minute out of every 10 minutes. ES will be delivered for up to 10 weeks or until the wound is healed for 3 days. The exciflex bandage will be changed when indicated clinically or every 5 days, whichever is sooner. At each bandage change, wound status monitored as described above, specifically a 3D digital image and wound swabs will be obtained. The exciflex power/control module will then be transferred to a new sterile flexible substrate and the exciflex bandage reapplied to the wound.
  Interventions: Device: exciflex
- Group B: Wound treated using standard of care (No Intervention): Control treated wounds in Group B participants will be covered with a standard of care hydrogel dressing such as Restore (Hollister Inc) together with Tegaderm . The SoC dressing will be used for up to 10 weeks or until the wound is healed for 3 days. The SoC bandage will be changed when indicated clinically or every 5 days, whichever is sooner. At each bandage change, wound status monitored as described above, specifically a 3D digital image and wound swabs will be obtained. A fresh sterile SoC bandage will then be reapplied to the wound.

INTERVENTIONS:
Device: exciflex — untethered electronic bandage with all the components of a surface stimulation system mounted on a flexible substrate.
  Arms: Group A: Wound treated using exciflex

SUMMARY:
Objectives: The study objective is to carry a pilot clinical assessment comparing the exciflex bandage to standard of care (SoC) for ischemic wounds and will involve participants who are Veterans with lower extremity ischemic wounds.

Research Plan: The study will employ a randomized repeated measures design to assess the therapeutic effectiveness of exciflex in clinical use.

Methodology: All participants with chronic ischemic wounds treated at LSCDVAMC will be potentially eligible for the study. Primary target populations will include Veterans with SCI who are inpatients or residents of the on-site Long Term Care Unit and Veterans with diabetes being followed by the Podiatry Service for wound care. In addition to meeting the general inclusion criteria noted above, further exclusion criteria relating to clinical factors include; (1)Age less than 18 years and (2)Pregnancy.

Clinical Significance: Chronic ischemic wounds fail to heal normally and are a major challenge in the long-term care of many Veterans. The exciflex bandage can improve outcomes and lower cost by automatically delivering electrotherapy without disturbing the wound dressing for up to seven days, unless indicated. The overall study goal is to complete pre-market testing and evaluation of the exciflex bandage system.

DETAILED DESCRIPTION:
The study will employ a randomized repeated measures design to assess the therapeutic effectiveness of the exciflex bandage in clinical use. Progressive changes in wound size, indicative of wound healing, will be determined using 3D digital stereophotogrammetry (LifeViz 3D system, Quantificare Inc., San Mateo, CA) together with wound swabs to collect wound bed fluid. The study cohort will comprise Veterans with ischemic wounds.

A parallel-group randomization will be used and participants will be randomly assigned to one of two groups: the experimental or investigation group (Group A) or the control group (Group B). Random allocation software will be used to produce qualified lists for parallel group assignment a priori and ensure that participants are randomized into groups that result in equal sample sizes Each will have a 50% chance of being assigned to either group. Group A will include eight (8) participants using the study device. Group B will include eight (8) participants undergoing standard of care treatment (SoC) with no study device.

ELIGIBILITY:
Inclusion Criteria:

* All participants with chronic ischemic wounds treated at LSCVAMC will be potentially eligible for the study
* Primary target populations will include Veterans with SCI who are inpatients or residents of the on-site Long-Term Care Unit and Veterans with diabetes being followed by the Podiatry Service for wound care

Exclusion Criteria:

In addition to meeting the general inclusion criteria noted above, further exclusion criteria relating to clinical factors include:

* Age less than 18 years.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Digital imaging | At each bandage change for up to 6 weeks
  Quantify wound size (mm2 for surface area, mmm3 for volume). The outcomes measures of wound surface area & wound volume are done by the investigators' 3D wound imaging camera that produces a digital output which includes both wound surface area (SA) & wound volume. One is derived from the other, i.e. Wound volume = SA x average depth.
IR imaging | At each bandage change for up to 6 weeks
  Wound bed temperature (degrees C)
Laser Speckle imaging | At each bandage change for up to 6 weeks
  Wound region blood flow (blood perfusion using arbitrary units)

SECONDARY OUTCOMES:
Wound swabs | At every bandage change for up to 6 weeks
  Further analysis using real-time polymerase chain reaction (PCR) for assessment of wound infection and healing biomarkers, including but not limited to VEGF and TNF-alpha. rt-PCR is a single assessment process to measure multiple biomarkers of wound infection and healing from a single sample, using plates that contain up to 96 different biomarkers each.

CONTACTS AND LOCATIONS:
Overall Officials: Kath M. Bogie, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No